CLINICAL TRIAL: NCT06494735
Title: Effect of the French Version If the Metagognitive Bibliotherapy Program "MYMCT" on Obsessive-compulsive Symptoms
Acronym: M-TOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-AOI-02
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyMCT Group (Experimental): Use of the bibliotherapy program
  Interventions: Behavioral: MyMCT
- Witness Group (No Intervention): Not using the bibliotherapy program

INTERVENTIONS:
Behavioral: MyMCT — Using the french version of the metagognitive bibliotherapy MyMCT
  Arms: MyMCT Group

SUMMARY:
Obsessive-compulsive disorder (OCD) is a psychiatric illness characterized by the presence of obsessions and/or compulsions. Without effective treatment, symptoms tend to worsen and become chronic. International guidelines recommend medication and/or psychotherapy as the first-line treatment for OCD. However, the majority of sufferers remain undertreated worldwide. This lack of access to care worsened during the Covid-19 pandemic. Much of this suffering could be avoided by facilitating access to evidence-based therapies. As such, many distance therapeutic interventions have recently developed, such as bibliotherapy. These unguided self-help programs are mostly based on approaches derived from cognitive behavioral therapies (CBTs). Specialized metacognition bibliotherapy is more specifically based on the hypothesis of a cognitive meta-level that affects off-line knowledge and on-line self-regulatory behaviors.

Yet, the majority of OCD sufferers are reported to exhibit inadequate metacognitive processing. Although these metacognitive abilities are often neglected in the OCD literature, they appear to play a significant causal role in the onset and maintenance of obsessive-compulsive symptoms. As a result, OCD-specific metacognitive treatments need to be developed to reduce symptomatology and improve quality of life for these patients. To date and to our knowledge, there is only one validated metacognitive bibliotherapeutic program for OCD. This manual is called "MyMCT: My MetaCognitive Training". A recent meta-analysis confirms its effectiveness with 373 participants from Germany, Switzerland and Russia in reducing obsessions and compulsions. Although these results are promising, MyMCT did not exist in a French version until 2021. Our team then translated the manual on a not-for-profit basis, and an independent translator at Nice University Hospital confirmed that it faithfully transcribed the meaning of the English version. This version has been freely available since November 2021 on the website of the Department of Psychiatry and Psychotherapy at Hamburg-Eppendorf University Medical Center (https://clinical-neuropsychology.de/metacognitive-training-for-ocd-mymct/).

The investigator propose to carry out a single-center randomized controlled research protocol concerning the effects of the French version of MyMCT in OCD patients. This clinical trial will be carried out́ in collaboration with Professor Moritz, author of MyMCT and renowned researcher.

ELIGIBILITY:
Inclusion Criteria:

* With OCD diagnosed by a psychiatrist,
* Unchanged psychiatric medication over the past 3 months,
* Have a good command of the French language,

Exclusion Criteria:

* Person with a psychotic or bipolar comorbidity diagnosed by a psychiatric physician
* Person participating simultaneously in another clinical trial interfering with the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | 2 month
  the intensity of obsessive-compulsive symptoms will be assessed using Yale Brown Obsessive Compulsive Scale (Y-BOCS). A global evaluation of symptoms (/40) is calculated using two subscores: 1. obsessions (/20); 2. compulsions (/20).

CONTACTS AND LOCATIONS:
Overall Officials: Bruno GIORDANA, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No